CLINICAL TRIAL: NCT07325357
Title: A Single-center, Randomized, Double-blind, Controlled Study Comparing the Efficacy and Safety of Pirfenidone Versus Placebo in the Treatment of Takayasu Arteritis on the Basis of Conventional Immunosuppressive Therapy
Brief Title: Effect of Pirfenidone on TA Fibrosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-Fibrosis with PFD
Record Dates: First submitted 2025-11-27; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Takayasu Arteritis
Keywords: fibrosis; pirfenidone; inflammation; Takayasu arteritis
MeSH Terms: conditions — Takayasu Arteritis; Fibrosis; Inflammation | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- pirfenidone (Experimental)
  Interventions: Drug: Pirfenidone Capsules

INTERVENTIONS:
Drug: Pirfenidone Capsules — pirfenidone 400mg.tid.po, escalated to 600mg.tid.po if acceptable in patients.
  Arms: pirfenidone
Drug: Placebo — Placebo capsules for pirfenidone.
  Arms: placebo

SUMMARY:
Takayasu arteritis is a severe vasculitis which could lead to significant disability and even death. While standard anti-inflammatory treatments can manage the systemic inflammation, they failed to stop a key driver of the disease: vascular fibrosis. This fibrosis could result in blood vessels thickening and narrowing, which continues to progress in many patients.

To tackle this critical treatment gap, the present project explores a new strategy. Building on pirfenidone's success in treating fibrosis in organs just like lungs and liver, along with promising early observations from our center, investigators believe adding this anti-fibrotic drug to standard therapy could improve vessel injury directly.

Therefore, investigators plan to conduct a clinical trial comparing pirfenidone with placebo in patients with Takayasu arteritis. The goal is to determine if this approach can successfully improve vascular injury and patient outcomes ultimately.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed the informed consents and meet the ACR 2022 classification criteria for Takayasu arteritis.
2. Male or female, age between 18 and 60 years.
3. Female patients must have a negative serum or urine pregnancy test and do not have pregnancy plans during the study period.
4. Within the 3 months prior to enrollment, the patient's treatment regimen must consist of glucocorticoids and immunosuppressants (methotrexate). Biological agents (IL-6R, TNF, or monoclonal antibody) might be used based on clinical need. Other targeted therapies (such as CD20 monoclonal antibodies, JAK inhibitors, etc.) or cell-based therapies (such as CAR-T or stem cell therapy) are not permitted.
5. During the 6-month follow-up period, the dosage and frequency of existing methotrexate and biologics (IL-6R monoclonal antibody, TNF monoclonal antibody, IL17 monoclonal antibody) must remain unchanged, except for adjustments of glucocorticoid doses based on clinical condition.
6. After 3 months of the above combination glucocorticoid and immunosuppressants, patients must achieve remission of disease activity (NIH score <2) and meet at least 3 of the following 5 criteria:

   i. Thickening of the affected vessel wall accompanied by luminal stenosis validated by angiographic examination.

ii. Carotid ultrasound showing medium-to-high echogenicity of the carotid artery wall.

iii. Progression in the thickness of the affected arterial wall compared to previous 3 months, with or without progression of luminal stenosis.

iv. Improvement in the thickness of the affected arterial wall of <10% compared to previous 3 months.

v. Within the 3 months prior to enrollment, the occurrence of new vascular ischemic symptoms or ischemic events, or worsening of pre-existing vascular ischemic symptoms. The ischemic symptoms or events must meet at least one of the criteria listed in the table below: Category (Criterion) Vascular Ischemic Signs

1. New emerged vascular bruits (carotid, subclavian, or renal arteries).
2. Newly emerged absent pulses (carotid, subclavian, brachial, radial, femoral, or dorsalis pedis arteries).
3. New emerged systolic blood pressure difference ≥10 mmHg between left and right arms.
4. New emerged systolic blood pressure difference ≥30 mmHg between ipsilateral upper and lower limbs.
5. Intermittent claudication in upper or lower limbs.

Cardiac

1. For non-hypertensive patients, blood pressure elevation to >140/90 mmHg.
2. For hypertensive patients, an increase in diastolic blood pressure ≥20 mmHg from baseline.
3. Ischemic angina.
4. Myocardial infarction.
5. Aortic valve insufficiency (moderate or severe).

Cerebral

1. Ischemic stroke.
2. New emerged ischemic symptoms: syncope, visual or auditory abnormalities such as decreased vision, visual field defects, etc.
3. CT cerebral perfusion imaging indicating ischemic or infarcted areas (with a corresponding volume >10 ml detected by CTP software).

Renal Radionuclide renogram showing a decrease in glomerular filtration rate over 10%; or an increase in serum creatinine exceeding 50% compared with the baseline.

Exclusion Criteria:

1. Presence of autoimmune diseases or autoinflammatory diseases other than Takayasu arteritis (e.g., systemic lupus erythematosus, ankylosing spondylitis, rheumatoid arthritis, etc.);
2. Use of antifibrotic drugs or drugs with potential antifibrotic properties (such as acetylcysteine, nintedanib, pirfenidone, etc.) within 6 months prior to enrollment, or participation in other clinical trials involving antifibrotic therapies;
3. Impaired liver function (elevated transaminases ALT/AST >2 times the upper limit of normal, or bilirubin exceeding the upper limit of normal), severe renal insufficiency (eGFR <15 mL/min/1.73m²), or requirement for psychotropic medications (excluding sleep medicine for sleep disorders);
4. Any severe, progressive, or uncontrolled concurrent hematological, gastrointestinal, pulmonary, cardiac, neurological, or other medical conditions unrelated to Takayasu arteritis which could pose unpredictable risks, in the investigator's judgment;
5. Allergy to the investigational drug or previous failure of regular pirfenidone treatment for 3 months;
6. Due to pirfenidone's metabolism primarily via cytochrome P450 isoenzymes (particularly CYP1A2), use of CYP1A2 inducers or inhibitors prior to enrollment must be discontinued and avoided throughout the study period; such medications are also prohibited during the study unless deemed medically necessary by the investigator for managing adverse events;
7. History of allergy to MRA contrast agents;
8. Planned vascular surgery during the 6-month follow-up period which may interfere with assessment results.

CYP1A2 Inhibitors:

Acyclovir, amiodarone, atazanavir, caffeine, cimetidine, ciprofloxacin, enoxacin, famotidine, flutamide, fluvoxamine, lidocaine, lomefloxacin, mexiletine, moclobemide, norfloxacin, ofloxacin, perphenazine, propafenone, ropinirole, tacrine, ticlopidine, tocainide, verapamil

CYP1A2 Inducers:

Carbamazepine, esomeprazole, griseofulvin, lansoprazole, moricizine, omeprazole, rifampin, ritonavir

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the effectiveness of pirfenidone in the treatment of Takayasu arteritis compared to the placebo | "From enrollment to the end of treatment at 6 months"
  Compared to placebo, the effectiveness of pirfenidone in the treatment of Takayasu arteritis is assessed with a composite endpoint. It indicates both clinical remission and imaging efficacy criterias must be met simultaneously, as follows:
  Clinical remission should meet all of the following criterias (①-④):
  * Absence of systemic symptoms such as fever, fatigue, or weight loss;
    * No new vascular symptoms or signs, and no worsening of pre-existing vascular symptoms; ③ No new ischemic symptoms or signs, and no worsening of pre-existing ischemic symptoms; ④ Normal erythrocyte sedimentation rate (if abnormal, non-disease activity factors must be excluded; a repeat test should be performed for evaluation);
  Note: If any of the following events occur in the CTCAE 5.0 grade increasing from baseline and reach grade 2 or higher, the case will be directly classified as not remission. These events include: ischemic stroke, syncope, intermittent claudication, and myocardial infarction.

SECONDARY OUTCOMES:
The radiographic response rate of pirfenidone in the treatment of Takayasu arteritis at 6th month, compared to placebo. | From enrollment to the end of treatment at 6 months
  1. Imaging Effective: Vascular ultrasound or MRA confirms a ≥30% reduction in the thickness of the affected vessel wall compared to baseline, along with a ≥10% increase in vessel diameter.
  2. Imaging Improvement: Vascular ultrasound or MRA confirms a <30% reduction in the thickness of the affected vessel wall compared to baseline, along with a <10% expansion of the stenotic vessel diameter compared to baseline.
  3. Imaging Ineffective: Vascular ultrasound or MRA confirms any of the following: an increase in the thickness of the affected vessel wall compared to baseline, OR no expansion of the stenotic vessel diameter compared to baseline, OR the occurrence of an ischemic event.
Compared to placebo, the clinical remission rate of pirfenidone at the end of 6th month in the treatment of Takayasu arteritis. | From enrollment to the end of treatment at 6 months
Compared to placebo, the average dose of glucocorticoid at the end of 6th month in pirfenidone, in the treatment of Takayasu arteritis. | From enrollment to the end of treatment at 6 months
Compared to placebo, the incidence of ischemic events within 6 months for pirfenidone in the treatment of Takayasu arteritis. | From enrollment to the end of treatment at 6 months
Compared to placebo, changes of fibrosis markers (MMP-1, MMP-3, MMPP-9, TIMP-1, etc.) for pirfenidone in the treatment of Takayasu arteritis at the end of 6 months. | From enrollment to the end of treatment at 6 months
Compared to placebo， the improvement of quality of life at the end of month 6 with pirfenidone in the treatment of Takayasu arteritis (assessed by SF-36). | From enrollment to the end of treatment at 6 months
  In the SF-36 scale, higher score indicates better outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma LY, Li CL, Chen RY, Dai XM, Ji ZF, Chen HY, Han H, Huang BJ, Sun Y, Jiang LD. The value of ultrasonography combined with clinical features for predicting carotid imaging progression of Takayasu's arteritis: a prospective cohort study. Clin Exp Rheumatol. 2021 Mar-Apr;39 Suppl 129(2):101-106. doi: 10.55563/clinexprheumatol/1o86of. Epub 2021 Mar 17. PMID 33734971
- [Background] Ma LY, Li CL, Ma LL, Cui XM, Dai XM, Sun Y, Chen HY, Huang BJ, Jiang LD. Value of contrast-enhanced ultrasonography of the carotid artery for evaluating disease activity in Takayasu arteritis. Arthritis Res Ther. 2019 Jan 16;21(1):24. doi: 10.1186/s13075-019-1813-2. PMID 30651132
- [Background] Lewis GA, Dodd S, Clayton D, Bedson E, Eccleson H, Schelbert EB, Naish JH, Jimenez BD, Williams SG, Cunnington C, Ahmed FZ, Cooper A, Rajavarma Viswesvaraiah, Russell S, McDonagh T, Williamson PR, Miller CA. Pirfenidone in heart failure with preserved ejection fraction: a randomized phase 2 trial. Nat Med. 2021 Aug;27(8):1477-1482. doi: 10.1038/s41591-021-01452-0. Epub 2021 Aug 12. PMID 34385704
- [Background] Munoz-Espinosa LE, Torre A, Cisneros L, Montalvo I, Male R, Mejia S, Aguilar JR, Lizardi J, Zuniga-Noriega J, Eugenia Icaza M, Gasca-Diaz F, Hernandez-Hernandez L, Cordero-Perez P, Chi L, Torres L, Rodriguez-Alvarez F, Tapia G, Poo JL. Noninvasive Evaluation of Prolonged-Release Pirfenidone in Compensated Liver Cirrhosis. ODISEA Study, a Randomised Trial. Liver Int. 2025 Jun;45(6):e70131. doi: 10.1111/liv.70131. PMID 40402087
- [Background] Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, King TE Jr, Lancaster L, Sahn SA, Szwarcberg J, Valeyre D, du Bois RM; CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011 May 21;377(9779):1760-9. doi: 10.1016/S0140-6736(11)60405-4. Epub 2011 May 13. PMID 21571362
- [Background] Shah PV, Balani P, Lopez AR, Nobleza CMN, Siddiqui M, Khan S. A Review of Pirfenidone as an Anti-Fibrotic in Idiopathic Pulmonary Fibrosis and Its Probable Role in Other Diseases. Cureus. 2021 Jan 4;13(1):e12482. doi: 10.7759/cureus.12482. PMID 33564498
- [Background] Kong X, Xu M, Cui X, Ma L, Cheng H, Hou J, Sun X, Ma L, Jiang L. Potential Role of Macrophage Phenotypes and CCL2 in the Pathogenesis of Takayasu Arteritis. Front Immunol. 2021 May 17;12:646516. doi: 10.3389/fimmu.2021.646516. eCollection 2021. PMID 34079541
- [Background] Rongyi C, Xiaojuan D, Jinghua W, Lingying M, Xiaomin D, Lili M, Huiyong C, Lindi J, Ying S. High level of serum complement 3 is a risk factor for vascular stenosis progression in TA patients receiving tocilizumab: a prospective observational study. Arthritis Res Ther. 2023 Aug 2;25(1):137. doi: 10.1186/s13075-023-03106-7. PMID 37533103
- [Background] Hellmich B, Agueda A, Monti S, Buttgereit F, de Boysson H, Brouwer E, Cassie R, Cid MC, Dasgupta B, Dejaco C, Hatemi G, Hollinger N, Mahr A, Mollan SP, Mukhtyar C, Ponte C, Salvarani C, Sivakumar R, Tian X, Tomasson G, Turesson C, Schmidt W, Villiger PM, Watts R, Young C, Luqmani RA. 2018 Update of the EULAR recommendations for the management of large vessel vasculitis. Ann Rheum Dis. 2020 Jan;79(1):19-30. doi: 10.1136/annrheumdis-2019-215672. Epub 2019 Jul 3. PMID 31270110
- [Background] Maz M, Chung SA, Abril A, Langford CA, Gorelik M, Guyatt G, Archer AM, Conn DL, Full KA, Grayson PC, Ibarra MF, Imundo LF, Kim S, Merkel PA, Rhee RL, Seo P, Stone JH, Sule S, Sundel RP, Vitobaldi OI, Warner A, Byram K, Dua AB, Husainat N, James KE, Kalot MA, Lin YC, Springer JM, Turgunbaev M, Villa-Forte A, Turner AS, Mustafa RA. 2021 American College of Rheumatology/Vasculitis Foundation Guideline for the Management of Giant Cell Arteritis and Takayasu Arteritis. Arthritis Rheumatol. 2021 Aug;73(8):1349-1365. doi: 10.1002/art.41774. Epub 2021 Jul 8. PMID 34235884
- [Background] Arnaud L, Haroche J, Mathian A, Gorochov G, Amoura Z. Pathogenesis of Takayasu's arteritis: a 2011 update. Autoimmun Rev. 2011 Nov;11(1):61-7. doi: 10.1016/j.autrev.2011.08.001. Epub 2011 Aug 9. PMID 21855656
- [Background] Park SJ, Kim HJ, Park H, Hann HJ, Kim KH, Han S, Kim Y, Ahn HS. Incidence, prevalence, mortality and causes of death in Takayasu Arteritis in Korea - A nationwide, population-based study. Int J Cardiol. 2017 May 15;235:100-104. doi: 10.1016/j.ijcard.2017.02.086. Epub 2017 Feb 22. PMID 28283361
- [Background] Wen D, Du X, Ma CS. Takayasu arteritis: diagnosis, treatment and prognosis. Int Rev Immunol. 2012 Dec;31(6):462-73. doi: 10.3109/08830185.2012.740105. PMID 23215768